CLINICAL TRIAL: NCT05761756
Title: Applied Physiology of Oxygen Toxicity: Mechanisms in Humans
Brief Title: Oxygen Toxicity: Mechanisms in Humans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00112396
Record Dates: First submitted 2023-02-06; First posted 2023-03-09 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Oxygen Toxicity; Hypercapnia; Seizures
MeSH Terms: conditions — Hypercapnia; Seizures | interventions — Caffeine; Methylphenidate; Carbon Dioxide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sleep Deprivation (Active Comparator): Effect of sleep deprivation on HCVR and arterial PCO2 during submersed rest and exercise at 98 fsw. Ten subjects will be tested before and after 24 hours of sleep deprivation. The order of sleep deprivation vs. control will be randomized. Measurements at 98 fsw will be obtained at rest and during 10 minutes of moderate exercise in thermoneutral (29-30°C) water.
  Interventions: Behavioral: Sleep Deprivation
- Caffeine (Experimental): Effect of caffeine and methylphenidate on HCVR and arterial PCO2 during submersed rest and exercise at 98 fsw. Twenty subjects will be similarly sleep-deprived, tested as above and then re-tested tested following oral administration of administration of either oral caffeine (N=10) or methylphenidate (N=10). Pre-dive caffeine will be administered 500 mg orally [59]. Pre-dive methylphenidate will be administered as a single dose of 5 mg [60]. The order of drug administration vs. control will be randomized. Measurements at 98 fsw will be obtained at rest and during 10 minutes of moderate exercise in thermoneutral (29-30°C) water. fNIRS will be used to assess cerebral oxygenation and regional blood volume.
  Interventions: Drug: Caffeine
- Methylphenidate (Experimental): Effect of caffeine and methylphenidate on HCVR and arterial PCO2 during submersed rest and exercise at 98 fsw. Twenty subjects will be similarly sleep-deprived, tested as above and then re-tested tested following oral administration of administration of either oral caffeine (N=10) or methylphenidate (N=10). Pre-dive caffeine will be administered 500 mg orally [59]. Pre-dive methylphenidate will be administered as a single dose of 5 mg [60]. The order of drug administration vs. control will be randomized. Measurements at 98 fsw will be obtained at rest and during 10 minutes of moderate exercise in thermoneutral (29-30°C) water. fNIRS will be used to assess cerebral oxygenation and regional blood volume.
  Interventions: Drug: Methylphenidate
- Carbon Dioxide Exposure (Experimental): Effect of simulated chronic CO2 exposure on HCVR and arterial PCO2 during submersed rest and exercise at 98 fsw. Ten subjects will be studied before and after induction of metabolic alkalosis as described above with daily oral administration of sodium bicarbonate. Oral bicarbonate to simulate hypercapnia exposure will seek to increase serum bicarbonate to 30 mM/L via daily oral intake of 6 teaspoons of NaHCO3 for five days. Subsequently, blood will be drawn and intake adjusted as necessary [61]. The order of alkalization vs. control will be randomized. Measurements at 98 fsw will be obtained at rest and during 10 minutes of moderate exercise in thermoneutral (29-30°C) water.
  Interventions: Drug: Carbon Dioxide

INTERVENTIONS:
Behavioral: Sleep Deprivation — 24 hours sleep deprivation
  Arms: Sleep Deprivation
Drug: Caffeine — Oral administration of caffeine
  Arms: Caffeine
Drug: Methylphenidate — Oral administration of methylphenidate
  Arms: Methylphenidate
Drug: Carbon Dioxide — Oral administration of sodium bicarbonate to simulate carbon dioxide exposure
  Arms: Carbon Dioxide Exposure

SUMMARY:
The goal of this clinical trial is to learn about the mechanisms of oxygen toxicity in scuba divers. The main questions it aims to answer are:

* How does the training of respiratory muscles affect oxygen toxicity?
* How do environmental factors, such as sleep deprivation, the ingestion of commonly utilized medications, and chronic exposure to carbon dioxide, impact the risk of oxygen toxicity?
* How does immersion in water affect the development of oxygen toxicity?

Participants will be asked to do the following:

* Undergo a basic screening exam composed of health history, vital signs, and some respiratory function tests
* Train their respiratory muscles at regular intervals
* Exercise on a cycle ergometer both in dry conditions and underwater/under pressure in the context of medication, sleep deprivation, or carbon dioxide exposure

Researchers will compare the performance of each subject before and after the possible interventions described above to see if there are changes in exercise performance, respiratory function, cerebral blood flow, and levels of gene expression.

ELIGIBILITY:
Inclusion Criteria:

* Equal numbers of male and female
* Non-smokers
* Aged 18-45 years
* Males will be required to have VO2 peak > or equal to mL/kg min
* and females > or equal to 30 mL/kg min

Exclusion Criteria:

* Pregnancy
* Cardiorespiratory disease, including hypertension
* Neuromuscular disease
* Anemia
* History of hemoglobinopathy, including sick cell disease and trait

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Hypercapnic ventilatory response | 3 months

SECONDARY OUTCOMES:
Lactate, pyruvate | 3 months
Arterial PCO2 | Baseline and after Intervention/arm
Integrated diaphragmatic function (IDF) composite score | Baseline and after Intervention/arm, which averages 3 months
  A composite score comprised of maximum breathing capacity (MBC), maximum inspiratory pressure (MIP), maximum expiratory pressure (MEP), and diaphragmatic thickness will be used as the measure of Integrated diaphragmatic function (IDF).
Cerebral blood oxygenation | Baseline and after Intervention/arm, which averages 3 months
Hormone levels (leptin, adiponectin) | Baseline and after Intervention/arm, which averages 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Derek B Covington, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health Sustem, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunworth SA, Natoli MJ, Cooter M, Cherry AD, Peacher DF, Potter JF, Wester TE, Freiberger JJ, Moon RE. Hypercapnia in diving: a review of CO(2) retention in submersed exercise at depth. Undersea Hyperb Med. 2017 May-Jun;44(3):191-209. doi: 10.22462/5.6.2017.1. PMID 28779577
- [Background] Drummond JC. Blood Pressure and the Brain: How Low Can You Go? Anesth Analg. 2019 Apr;128(4):759-771. doi: 10.1213/ANE.0000000000004034. PMID 30883421
- [Background] Lucas SJ, Tzeng YC, Galvin SD, Thomas KN, Ogoh S, Ainslie PN. Influence of changes in blood pressure on cerebral perfusion and oxygenation. Hypertension. 2010 Mar;55(3):698-705. doi: 10.1161/HYPERTENSIONAHA.109.146290. Epub 2010 Jan 18. PMID 20083726
- [Background] Wester TE, Cherry AD, Pollock NW, Freiberger JJ, Natoli MJ, Schinazi EA, Doar PO, Boso AE, Alford EL, Walker AJ, Uguccioni DM, Kernagis D, Moon RE. Effects of head and body cooling on hemodynamics during immersed prone exercise at 1 ATA. J Appl Physiol (1985). 2009 Feb;106(2):691-700. doi: 10.1152/japplphysiol.91237.2008. Epub 2008 Nov 20. PMID 19023017
- [Background] Pendergast DR, Moon RE, Krasney JJ, Held HE, Zamparo P. Human Physiology in an Aquatic Environment. Compr Physiol. 2015 Sep 20;5(4):1705-50. doi: 10.1002/cphy.c140018. PMID 26426465
- [Background] Linnarsson D, Ostlund A, Lind F, Hesser CM. Hyperbaric bradycardia and hypoventilation in exercising men: effects of ambient pressure and breathing gas. J Appl Physiol (1985). 1999 Oct;87(4):1428-32. doi: 10.1152/jappl.1999.87.4.1428. PMID 10517774
- [Background] Oppersma E, Doorduin J, van der Hoeven JG, Veltink PH, van Hees HWH, Heunks LMA. The effect of metabolic alkalosis on the ventilatory response in healthy subjects. Respir Physiol Neurobiol. 2018 Feb;249:47-53. doi: 10.1016/j.resp.2018.01.002. Epub 2018 Jan 4. PMID 29307724
- [Background] Cherry AD, Forkner IF, Frederick HJ, Natoli MJ, Schinazi EA, Longphre JP, Conard JL, White WD, Freiberger JJ, Stolp BW, Pollock NW, Doar PO, Boso AE, Alford EL, Walker AJ, Ma AC, Rhodes MA, Moon RE. Predictors of increased PaCO2 during immersed prone exercise at 4.7 ATA. J Appl Physiol (1985). 2009 Jan;106(1):316-25. doi: 10.1152/japplphysiol.00885.2007. Epub 2008 Sep 11. PMID 18787095
- [Background] Dodson ME, Fryer JM. Postoperative effects of methylphenidate. Br J Anaesth. 1980 Dec;52(12):1265-70. doi: 10.1093/bja/52.12.1265. PMID 7004471
- [Background] GALE AS. The effect of methylphenidate (ritalin) on thiopental recovery. Anesthesiology. 1958 Jul-Aug;19(4):521-31. doi: 10.1097/00000542-195807000-00009. No abstract available. PMID 13545587
- [Background] Beecroft J, Duffin J, Pierratos A, Chan CT, McFarlane P, Hanly PJ. Enhanced chemo-responsiveness in patients with sleep apnoea and end-stage renal disease. Eur Respir J. 2006 Jul;28(1):151-8. doi: 10.1183/09031936.06.00075405. Epub 2006 Mar 1. PMID 16510459
- [Background] Yao Q, Pho H, Kirkness J, Ladenheim EE, Bi S, Moran TH, Fuller DD, Schwartz AR, Polotsky VY. Localizing Effects of Leptin on Upper Airway and Respiratory Control during Sleep. Sleep. 2016 May 1;39(5):1097-106. doi: 10.5665/sleep.5762. PMID 26951402
- [Background] Eynan M, Arieli Y, Taran B, Yanir Y. Symptoms of central nervous system oxygen toxicity during 100% oxygen breathing at normobaric pressure with increasing inspired levels of carbon dioxide: a case report. Diving Hyperb Med. 2020 Mar 31;50(1):70-74. doi: 10.28920/dhm50.1.70-74. PMID 32187621
- [Background] Martin BJ. Effect of sleep deprivation on tolerance of prolonged exercise. Eur J Appl Physiol Occup Physiol. 1981;47(4):345-54. doi: 10.1007/BF02332962. PMID 7199438